CLINICAL TRIAL: NCT04249479
Title: The Effect of ContrAst Media Temperature on Patient Comfort in Computed tomograpHY of the Abdomen.
Brief Title: Contrast Media Temperature and Patient Comfort in CT of the Abdomen
Acronym: CATCHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NL68789.068.19
Record Dates: First submitted 2019-12-01; First posted 2020-01-31 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Contrast Media; Comfort; Temperature; Abdomen
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Intervention Model Description: It is a double-blinded randomised controlled non-inferiority trial conducted according to Guidelines of Good Clinical Practice. The aim of the study is to prospectively compare room temperature CM to pre-warmed CM with regard to image quality, safety, and participant comfort in portal venous abdominal imaging.
  We are aiming to prospectively enrol 216 consecutive patients, who will be scheduled for contrast enhanced abdominal CT.
  216 patients will be divided into 2 different groups:
  * Group I: 300 mg/ml at a temperature of 20° C
  * Group II: 300 mg/ml at a temperature of 37° C Iodine concentrated CM of 300 mg/ml is clinically used as a standard routine injection protocol for all CT scans in our department, including abdominal CT. The scan protocol is identical to our daily clinical practice. The only difference is that 50% of the included patients will receive CM warmed at room temperature. Both CM temperatures are saved/warmed in an incubator.
Who Masked: Participant, Investigator
Masking Description: All subjects will be randomized into two different groups as listed in the study outline.
  The randomization schedule will be prepared and centrally administered. A computer random number generator prepares the randomization schedule in a 1:1 fashion (balanced randomization). Stratification is performed, based on age (< 60 and ≥ 60 years) and weight (< 80 and ≥ 80 kg). Variable block randomization will distribute patients equally over time.
  The blinding and randomization process will be conducted by Clinical Trial Centre Maastricht (CTCM, www.CTCM.nl) with a randomization program designed for usage of different techniques (minimization, block method, biased-coin, etc). The technician who administers the CM is aware of the CM temperature. Therefore, the technicians will be instructed before start of the study, not to give this information to the patient, not even when requested by the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM temperature 20° C (Experimental): CM is administered to the patient at a temperature of 20° C.
  Interventions: Other: CM Temperature (20° C); Other: Weight
- CM temperature 37° C (Active Comparator): CM is administered to the patient at a temperature of 37° C.
  Interventions: Other: CM Temperature (37° C); Other: Weight

INTERVENTIONS:
Other: CM Temperature (20° C) — CM will be administered at 20° C (room temperature).
  Arms: CM temperature 20° C
Other: CM Temperature (37° C) — CM will be administered at 37° C (pre-heated).
  Arms: CM temperature 37° C
Other: Weight — The patients' weight is measured prior to scanning by a technician on a weighing scale available in the scanner room.

SUMMARY:
Abdominal computed tomographic (CT) is an important prognostic tool with regard to the detection of oncological, infectious and other abdominal disorders.

The total iodine load (TIL) is regarded as a decisive factor in the opacification of parenchymal structures. The EICAR trial demonstrated that injection with high flow rates of prewarmed contrast media (CM) was safe and patients did not experience any pain, stress of discomfort during injection. Flow rates as high as 8.8 ml/s were injected without any discomfort. All concentrations used (e.g. 240, 300 and 370 mg I/ml) in this study were prewarmed. According to the recent recommendations (ESUR guidelines 10.0) it should be considered to warm iodine-based CM before administration. The hypothesis is that although using CM at room temperature (~23°C [~73°F]) might result in lower attenuation of the liver parenchyma than would be achieved using CM pre-warmed to body temperature, diagnostic image quality, patient safety and comfort will not be compromised by not pre-warming CM in this setting. According to the guidelines, it is regarded as best clinical practice to pre-warm CM. Surprisingly, these recommendations are merely based on a hypothetical assumption. In the literature, there are no studies evaluating this topic and it has never been clearly shown to result in a better patient comfort. For this reason, many clinics do not pre-warm their CM in daily clinical routine. Only one study evaluated subjective comfort in hysterosalpingography (HSG), in which CM is injected in to the cavity of the uterus. This study found that prewarmed CM alleviates the pain and decreased the incidence of vasovagal episodes during HSG. To the best of our knowledge, no study showed that prewarmed CM in CT resulted in higher patient comfort, in comparison to CM at room temperature (20° C).

Up till now, all CM in the department is prewarmed. In case this study does not show a difference in patient comfort, prewarming the CM can be stopped, resulting in a considerable simplified workflow.

The hypothesis is that usage of CM at room temperature (20° C) might result in a decreased level of patient comfort in abdominal CT, in comparison to pre-heated (37° C) CM, with no significant difference in diagnostic attenuation of the liver parenchyma between groups.

DETAILED DESCRIPTION:
Abdominal computed tomography (CT) scans are performed daily on a regular basis. Since its advent, rapid technical advances in CT continuously improved image quality. Besides scan technique, the contrast media (CM) injection protocol is the crucial factor in abdominal imaging. Parenchymal contrast enhancement is determined by patient related factors (e.g. cardiac output, blood volume and patient weight), the CM injection protocol and the scan protocol. Much literature has been performed with regard to optimizing CM application and the scan protocol. Flow rate of the CM and patient discomfort have been thoroughly investigated in our department. Heating CM up to body temperature has been daily clinical routine in our department for years.

According to the recent recommendations (ESUR guidelines 10.0) it is advised to warm iodine-based CM before administration. Warming the CM is expected to result in a higher patient comfort, based on clinical observation. Kok et al. showed in phantom experiments that high temperature, low iodine concentration and low viscosity significantly decreases injection pressure. Subsequently, as increased temperature reduces the viscosity of the CM, the decreased viscosity is hypothesized to reduce the risk of extravasation. A decreased viscosity might also have a substantial impact on individual tailored CM injection protocols in daily routine scanning as it is speculated that a decrease of viscosity and subsequent decrease in peak injection pressure could influence patient comfort during injection. The EICAR trial showed that prewarmed CM can be safely injected at high flow rates, without patient discomfort, pain or stress. However, the latter was not compared to CM at room temperature.

Different CM concentrations are used in different hospitals throughout the world. The higher the concentration, the higher the viscosity of the CM. In present study, only one CM concentrations (e.g. 300 mg/ml) will be used, which is used in daily clinical practice for years. Heating the CM decreases the viscosity. It is therefore expected that the preheated CM in a concentration of 300 mg/ml has a lower viscosity in comparison to the CM at 20° C.

Pre-warming CM might be regarded as best clinical practice. No studies have been performed to investigate this statement, nor is there any literature that shows that prewarmed CM has a favorable patient comfort compared to CM injected at room temperature. For these reasons, there remains to be some reluctance and many clinics still not pre-warm their CM. One study, in which CM is injected in to the cavity of the uterus to check for any anatomical variants and causes for infertility, showed a preference for prewarmed CM in hysterosalpingography (HCG). This study found that prewarmed CM alleviates the pain and decreased the incidence of vasovagal episode during the HCG.

The hypothesis is that although using CM at room temperature (~23°C [~73°F]) might result in lower attenuation of the liver parenchyma than would be achieved using CM pre-warmed to body temperature, diagnostic image quality, patient safety and comfort will not be compromised by not pre-warming CM in this setting. Pre-warming CM requires special equipment and more complex planning and logistics. On the other hand, pre-warming CM may yield higher attenuation levels, comfort and image quality. In case this study does not show a significant difference in patient comfort and diagnostic quality between groups, pre-warming the CM can be stopped, resulting in a considerable simplified workflow.

ELIGIBILITY:
Inclusion criteria

* Patients referred for abdominal CT
* Patient ≥ 18 years old and competent to sign informed consent

Exclusion criteria

* Hemodynamic instability
* Pregnancy
* Renal insufficiency defined as glomerular filtration rate (GFR) < 30ml/min/1.73m2 (Odin protocol 004720)
* Iodine allergy (Odin protocol 022199)
* Age < 18 year
* Unable to give informed consent or no informed consent obtained
* Inability to position an 18 gauge cannula in an antecubital vein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Liver attenuation | Expected within one month after the CT is performed
  Mean attenuation in Hounsfield Units (HU) is based on three liver segments, preferably segments 2, 5 and 8 (Couinaud classification). Absolute difference in mean attenuation of the liver parenchyma between groups was calculated with a two-sided 95% confidence interval of the difference.

SECONDARY OUTCOMES:
Patient comfort | Immediately after CT
  Patient (dis)comfort during and after injection of CM with varying temperatures, rated on a questionnaire
Pain during injection | Questionnaire immediately after CT
  Assessed with a questionnaire with the option yes/no
Pain rate | Questionnaire immediately after CT
  Assessed with a 11-point numeric rating scale (0=no pain; 10=very severe pain)
Different physiological reactions and sensations injection | Immediately after the CT
  Questionnaire has to be filled in which people can tick a box if they had feelings of shivering/goosebumps/or being cold. There is some free space to write down other sensations.
Objective image quality - Signal-to-noise ratio | Within one month after the CT is performed
  mean attenuation of the liver divided by the mean standard deviation
Objective image quality - Contrast-to-noise ratio | Within one month after the CT is performed
  Mean liver attenuation minus HU of the left paraspinal muscle, divided by the SD of the attenuation of the paraspinal muscle
Subjective image quality | Within one month after the end of the study
  Rated in consensus on a 5-point Likert scale by two readers
Body weight | Right before the scan is performed
  Weight is measured on a weighing scale
CM volume | Information is expected to be collected from the Certegra form available in Impax within 1 month
  The milliliter of CM administered
Flow rate | Information is expected to be collected from the Certegra form available in Impax within 1 month
  Flow rate of the contrast media in ml/s
Injection site | Information is expected to be collected from the Certegra form available in Impax within 1 month
  Injection site of the CM
Catheter Gauge | Information is expected to be collected from the Certegra form available in Impax within 1 month
  Catheter size used for CM injection
Effective milliamperes (mAs) | Information is expected to be collected from the Certegra form available in Impax within 1 month
  The effective mAs used in the specific patient
CT Dose Index (CTDI)vol | Information is expected to be collected from Impax within 1 month
  CTDIvol (in mGy) the patient received
Dose-length product (DLP) | Information is expected to be collected from Impax within 1 month
  DLP (in mGycm) the patient received
Tube voltage | Information is expected to be collected from Impax within 1 month
  Tube voltage used in the specific scan

CONTACTS AND LOCATIONS:
Overall Officials: Joachim E Wildberger, Professor, Principal Investigator — Maastricht University Medical Center
Locations (1):
- MaastrichtUMC, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The results will be published in international peer reviewed journals in order to spread new insights regarding contrast media temperature in abdominal CT imaging. Both positive and negative results will be published according to the guidelines of the 'Centrale Commissie Mensgebonden Onderzoek' (CCMO).
Supporting Information: CSR
Time Frame: Within 18 months after completion

REFERENCES:
- [Derived] Martens B, Wildberger JE, Van Kuijk SMJ, De Vos-Geelen J, Jeukens CRLPN, Mihl C. Influence of Contrast Material Temperature on Patient Comfort and Image Quality in Computed Tomography of the Abdomen: A Randomized Controlled Trial. Invest Radiol. 2022 Feb 1;57(2):85-89. doi: 10.1097/RLI.0000000000000807. PMID 34280944